CLINICAL TRIAL: NCT05755308
Title: Faecal Microbiota Transplantation to Ameliorate Nintedanib-induced Diarrhea in Patients With Idiopathic Pulmonary Fibrosis
Acronym: BIOFEV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RICHELDI LUCA, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5260
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Faecal microbiota transplantation (Experimental)
  Interventions: Procedure: Autologous FMT
- Placebo arm (Placebo Comparator)
  Interventions: Procedure: Placebo FMT

INTERVENTIONS:
Procedure: Autologous FMT — Autologous faecal microbiota transplantation by colonoscopy.
  Arms: Faecal microbiota transplantation
Procedure: Placebo FMT — Placebo FMT will consist of 250 mL water. Placebo infusions will be delivered by colonoscopy.
  Arms: Placebo arm

SUMMARY:
This is a multicentric, randomised, double-blind, placebo-controlled study that will consist of two consecutive phases:

1. First phase: faecal samples will be collected in patients diagnosed with Idiopathic pulmonary fibrosis treated with nintedanib.
2. Second phase: double-blind, randomised, clinical trial of autologous faecal microbiota transplantation (FMT) vs placebo in Idiopathic pulmonary fibrosis patients who will experience nintedanib-induced diarrhea within 8 weeks of baseline visit.

Follow-up visits will be scheduled at 1, 4 and 12 weeks after randomization. The main aim of the study is to assess the efficacy of FMT in ameliorating diarrhea experienced by patients with idiopathic pulmonary fibrosis treated with nintedanib.

ELIGIBILITY:
Inclusion Criteria:

Phase 1 (faecal samples collection)

* Patients aged ≥18 years when signing the informed consent;
* Diagnosis of IPF within 4 weeks based on 2018 ATS/ERS/JRS/ALAT Guidelines (2) as confirmed by the investigator based on chest HRCT scan and if available surgical lung biopsy;
* Patients already on antifibrotic therapy with nintedanib according to clinical practice.

Phase 2 (FMT procedure)

- Patients who develop diarrhea of grade 2 or 3 according to the Common Terminology Criteria (CTC) for Adverse Events (AE) version 5.0 (12) within 8 weeks of baseline visit.

Exclusion Criteria:

* Women of childbearing potential or pregnant;
* History of colorectal surgery or cutaneous stoma;
* Food allergies;
* Recent (<6 weeks) therapy with drugs that could possibly alter gut microbiota (e.g. antibiotics, probiotics, proton pump inhibitors, immunosuppressants and/or metformin);
* Any documented active or suspected malignancy, except appropriately treated basal cell carcinoma of the skin, "under surveillance" prostate cancer or in situ carcinoma of uterine cervix;
* Decompensated heart failure or heart disease with ejection fraction lower than 30%, severe respiratory failure, psychiatric disorders, pregnancy or inability to provide informed consent.
* Fecal sample unable for FMT according to the opinion of the Investigators (e.g. positive for pathogens);
* (phase 2 only) Diarrhea from known causes (e.g. infectious gastroenteritis, Clostridium difficile infection, coeliac disease, inflammatory bowel disease, irritable bowel syndrome, chronic pancreatitis and/or biliary salt diarrhea).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Resolution of diarrhea | 4 weeks
  Resolution of diarrhea at 4 weeks from FMT procedures.

SECONDARY OUTCOMES:
Number of Participants with Resolution of diarrhea | 1 and 12 weeks
  Resolution of diarrhea at 1 and 12 weeks from FMT procedures
Nintedanib discontinuation | 12 weeks
  Rate of nintedanib discontinuation or dose reduction
Intestinal microbiota composition | 1, 4 and 12 weeks
  Analysis of intestinal microbiota composition at baseline and at 1, 4 and 12 weeks after the end of FMT procedures
Forced vital capacity (FVC) | 12 weeks
  Relative and absolute change in forced vital capacity (FVC) percent-predicted from baseline at week 12
St. George's Respiratory Questionnaire (SGRQ) | 12 weeks
  Change in St. George's Respiratory Questionnaire (SGRQ) score from baseline at week 12
Exacerbation | 12 weeks
  Time to first acute exacerbation.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Roma, Italy